CLINICAL TRIAL: NCT07247513
Title: Glycaemic Responses to a Food Intake Sequence Intervention Under Free-living Conditions in Elite Female Athletes
Brief Title: Glycaemic Responses to a Food Intake Sequence Intervention in Free-living Elite Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Federação Portuguesa de Futebol (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FOODSEQ-GRFA; 2022.12954.BD (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Nutrition; Glycemic Variability; Dietary Intervention; Sleep; Exercise
Keywords: food order; meal sequence; glycaemia; sport nutrition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This trial is designed as a randomised, counterbalanced, crossover, open label, superiority trial with two groups. Block randomization will be performed by an external researcher with a 1:1 allocation ratio, and allocation concealment will be ensured through the use of sequentially numbered, opaque, sealed envelopes.
Masking Description: It is not possible to blind participants or researchers envolved in data collection to the intervention assigned in each period due to the nature of the intervention and comparator (food intake sequence of the same elements within a meal). However, both will be blinded to CGM data throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CL - CF (Experimental): The interventions (carbohydrate-last meal pattern (CL) or carbohydrate-first meal pattern (CF)) will be delivered in random order. If participants are allocated to this study arm, they will receive the CL on the first 2 days and the CF on the next 2 days of the study period.
  Interventions: Other: Carbohydrate-last meal pattern; Other: Carbohydrate-first meal pattern
- CF - CL (Active Comparator): The interventions (carbohydrate-last meal pattern (CL) or carbohydrate-first meal pattern (CF)) will be delivered in random order. If participants are allocated to this study arm, they will receive the CF on the first 2 days and the CL on the next 2 days of the study period.
  Interventions: Other: Carbohydrate-last meal pattern; Other: Carbohydrate-first meal pattern

INTERVENTIONS:
Other: Carbohydrate-last meal pattern — Participants will consume the main dietary sources of protein, fat, fibre and/or polyphenols before the main dietary sources of simple carbohydrate in the standardised test-meals (breakfast and supper) and will be encouraged to maintain this food intake sequence in the remaining meals of the day.
  Participants will be instructed to consume lunch and dinner within 30 min, and breakfast and supper within 15 min at a comfortable pace, without intervals between the carbohydrate and non-carbohydrate-rich meal components.
  Other Names: CL; CHO-last
Other: Carbohydrate-first meal pattern — Participants will consume the main dietary sources of protein, fat, fibre and/or polyphenols after the main dietary sources of simple carbohydrate in the standardised test-meals (breakfast and supper) and will be encouraged to maintain this food intake sequence in the remaining meals of the day.
  Participants will be instructed to consume lunch and dinner within 30 min, and breakfast and supper within 15 min at a comfortable pace, without intervals between the carbohydrate and non-carbohydrate-rich meal components.
  Other Names: CF; CHO-first

SUMMARY:
The goal of this clinical trial is to investigate the impact of a food intake sequence intervention under free-living conditions on glycaemic responses in elite female athletes. Specifically, the main questions it aims to answer are:

1. Does consuming breakfast in different food intake sequences alter postprandial interstitial glucose responses?
2. Does consuming a pre-exercise meal in different food intake sequences alter interstitial glucose responses during exercise?
3. Does consuming the last meal of the day in different food intake sequences alter nocturnal interstitial glucose responses?

To address these questions, researchers will compare eating the dietary sources of rapidly absorbed carbohydrate (CHO) at the end (CHO-last meal pattern) or at the start (CHO-first meal pattern) of standardised mixed meals, at different times of day, in a randomised, counterbalanced, crossover design.

Participants will wear a blinded continuous glucose monitor (CGM) for 6 consecutive days during a training camp. Throughout the study, they will be provided with buffet meals, at the same time and location each day. Dietary intake will be ad libitum, except for breakfast and supper, for which participants will select a preferred composition (ingredients, preparation methods, portion sizes) to replicate across study days. In all ad libitum meals (i.e., lunch, snacks, and dinner), they will be asked to maintain their assigned food intake sequence.

* On day 1, athletes will eat freely. An educational session on the study protocol and food sequence manipulation will be delivered, and informed consent, questionnaires, screening assessments, and CGM fitting will be completed. Data collected by the CGM during the first 24 hours will be disregarded due to sensor stabilisation. Hence, this period will serve for familiarisation only.
* On days 2 and 3, one group will eat the last meal of the day (i.e., supper) in a CHO-last meal pattern, while the other will follow a CHO-first meal pattern; on days 3 and 4 one group will eat breakfast in a CHO-last meal pattern while the other will follow a CHO-first meal pattern.
* On days 4 and 5 (supper) and 5 and 6 (breakfast), participants in each group will adhere to the alternate condition.

Concurrent data on potential confounding factors (e.g., dietary intake, physical activity, internal and external load during training sessions/competition, sleep quantity and quality, menstrual cycle phase/status) will be collected.

Due to the short camp duration, implementing a one-day washout period will not be feasible. Therefore, repeated measurements over two consecutive days per condition will be obtained to minimise carryover effects of the food intake sequence from prior meals on end-of-intervention data (the final 24 hours per condition), and to assess intraindividual consistency of outcomes at matched-times and standardised settings.

Glycaemic responses will be compared within-participant between food intake sequences using linear mixed models with random intercepts, to account for repeated measures, interindividual variability, and potential missing data.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-64 years old)
* Women
* Elite athletes (meeting training and performance caliber criteria ≥Tier 4; McKay et al., 2022)
* Healthy (meeting the exclusion criteria for medical conditions)
* Normal glucose tolerant according to the latest review standards of the American Diabetes Association (ElSayed et al., 2024): HbA1c <5.7%, fasting plasma glucose <5.6 mmol/L (100 mg/dL), or 2-h plasma glucose <7.8 mmol/L (140 mg/dL) during a 75-g OGTT
* Able and willing to provide informed consent and safely comply with study procedures

Exclusion Criteria:

* Any medical condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias into the experiment (e.g. pregnancy, alcohol or substance abuse; any condition affecting the glucose and lipid metabolism or appetite, reviewed on a case by case basis)
* Any reported medication or supplementation that may interfere with the glucose metabolism (e.g., acarbose, aspirin, berberine, insulin, metformin, semaglutide, sulfonylureas, thiazide diuretics, thiazolidinediones, vitamin C). Other medication and supplementation will be reviewed on a case by case basis.
* Recent change in body mass (± 2 kg in the last 2 months)
* Smoking

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender
Enrollment: 22 (Actual)
Dates: Start 2025-11-24 (Actual); Primary Completion 2025-11-29 (Actual); Study Completion 2025-11-29 (Actual)

PRIMARY OUTCOMES:
Incremental interstitial glucose peak after a standardised test meal | 0-120 minutes following a standardised test meal
  Difference between CHO-last and CHO-first meal patterns in the incremental interstitial glucose peak (mmol/L) adjusted for baseline, following standardised breakfasts (independent of and coinciding with subsequent exercise) and the end-of-intervention (days 3 and 5) standardised supper, assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ).

SECONDARY OUTCOMES:
Incremental area under the interstitial glucose curve after a standardised test meal | 0-120 minutes following a standardised test meal
  Difference between CHO-last and CHO-first meal patterns in the incremental area under the interstitial glucose curve (mmol/L x min) adjusted for baseline, following standardised breakfasts (independent of and coinciding with subsequent exercise) and the end-of-intervention (days 3 and 5) standardised supper, assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ).
Time-to-peak interstitial glucose after a standardised test meal | 0-120 minutes following a standardised test meal
  Difference between CHO-last and CHO-first meal patterns in the time-to-peak interstitial glucose (minutes), following standardised breakfasts (independent of and coinciding with subsequent exercise) and the end-of-intervention (days 3 and 5) standardised supper, assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ).
Time out of interstitial glucose range after a standardised test meal | 0-180 minutes following a standardised test meal
  Difference between CHO-last and CHO-first meal patterns in the time spent >7.8 mmol/L and time <3.9 mmol/L (%), following standardised breakfasts (independent of and coinciding with subsequent exercise) and the end-of-intervention (days 3 and 5) standardised supper, assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ).
Interstitial glucose dip after a standardised test meal | 0-180 minutes following a standardised test meal
  Difference between CHO-last and CHO-first meal patterns in the 2-3-hour interstitial glucose dip (mmol/L), following standardised breakfasts not coinciding with subsequent exercise, and the end-of-intervention (days 3 and 5) standardised supper, assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ).
Interstitial glucose concentrations during specific activities | 24 hours
  Difference between CHO-last and CHO-first meal patterns in the mean interstitial glucose concentrations (mmol/L) across 15-minute averages and adjusted for baseline where relevant, during the following periods: after standardised breakfasts (independent of and coinciding with exercise); after the end-of-intervention (days 3 and 5) standardised supper, during exercise not coinciding with postprandial periods, during evening sleep, and during daytime rest, assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ).
Within-day standard deviation of interstitial glucose | 24 hours
  Difference between CHO-last and CHO-first meal patterns in the 24-hour standard deviation (SD) of interstitial glucose concentrations during the end-of-intervention monitoring period (days 3 and 5), assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ sensor).
Within-day coefficient of variation of interstitial glucose | 24 hours
  Difference between CHO-last and CHO-first meal patterns in the 24-hour coefficient of variation (%) of interstitial glucose concentrations during the end-of-intervention monitoring period (days 3 and 5), assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ sensor).
Mean amplitude of glycaemic excursions (MAGE) | 24 hours
  Difference between CHO-last and CHO-first meal patterns in the mean amplitude of glycaemic excursions (MAGE) during the end-of-intervention monitoring period (days 3 and 5), assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ sensor).
Large amplitude of glycaemic excursions (LAGE) | 24 hours
  Difference between CHO-last and CHO-first meal patterns in the large amplitude of glycaemic excursions (LAGE) during the end-of-intervention monitoring period (days 3 and 5), assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ sensor).
Within-day time out of interstitial glucose range | 24 hours
  Difference between CHO-last and CHO-first meal patterns in the time spent >7.8 mmol/L and <3.9 mmol/L (%) over 24 hours during the end-of-intervention monitoring period (days 3 and 5), assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ sensor).
Between-day glycaemic variability | 24 hours
  Difference between CHO-last and CHO-first meal patterns in the mean of daily differences (MODD) of interstitial glucose responses at matched clock times, assessed using a blinded continuous glucose monitoring system (Freestyle Libre Pro IQ).

CONTACTS AND LOCATIONS:
Overall Officials: Rita Giro, Principal Investigator — Faculty of Nutrition and Food Sciences of the University of Porto (FCNAUP); FPF Academy, Federação Portuguesa de Futebol
Locations (1):
- Cidade do Futebol, Oeiras, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Anonymised IPD will be made available upon reasonable request directed to the corresponding author.
Supporting Information: SAP, ICF
Time Frame: IPD will become accessible following the publication of all study findings.
Access Criteria: IPD will be made available to researchers with legitimate scientific purposes (such as systematic reviews or meta-analyses).